CLINICAL TRIAL: NCT06231264
Title: A Multicenter Randomized Controlled Trial of Transcutaneous Electrical Acustimulation in the Treatment of Mild to Moderate Ulcerative Colitis
Brief Title: Transcutaneous Electrical Acustimulation in the Treatment of Mild to Moderate Ulcerative Colitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20232371
Record Dates: First submitted 2024-01-10; First posted 2024-01-30 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment group (Experimental): Subjects will be trained to use the devices at the treatment sites and receive treatment twice a day for 8 weeks.
  Interventions: Device: transcutaneous electrical acustimulation at treatment sites
- shame group (Placebo Comparator): Subjects will be trained to use the devices at the sham sites and receive sham treatment twice a day for 8 weeks.
  Interventions: Device: transcutaneous electrical acustimulation at sham sites

INTERVENTIONS:
Device: transcutaneous electrical acustimulation at treatment sites — A transcutaneous electrical stimulator (TEA) device applies a mild electric stimulation through the skin, similar to acupuncture at the treatment site. The precise stimulating sites are not described upon registration to reduce unblinding risk.
  Other Names: TEA
  Arms: treatment group
Device: transcutaneous electrical acustimulation at sham sites — A transcutaneous electrical stimulator (TEA) device applies a mild electric stimulation through the skin, similar to acupuncture at the sham treatment sites. The precise stimulating sites are not described upon registration to reduce unblinding risk.
  Other Names: sham-TEA
  Arms: shame group

SUMMARY:
The aim of this study was to evaluate the efficacy and safety of transcutaneous electrical acustimulation in patients with mild to moderate ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Ulcerative colitis diagnosed for at least 3 mouths.
3. Mayo score 4-10, Mayo endoscopic score 2-3 points
4. Resistant to at least one type of medical treatments

Exclusion Criteria:

1. Treatment-naive ulcerative colitis (no previous treatment)
2. Acute severe ulcerative colitis
3. Previous surgical treatment or severe colitis at imminent risk of surgery infective colitis
4. Other systemic diseases
5. Pregnancy and lactation
6. Allergic to the electrode patch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Clinical response | 8 weeks
  decrease of ≥3 points and ≥30% from baseline mayo score and decrease of ≥1 point in rectal bleeding subscore or absolute rectal bleeding subscore ≤ 1

SECONDARY OUTCOMES:
Change from baseline in the Mayo score | 8 weeks
  Mayo score at 8 week minus the Mayo score at baseline. The range of Mayo score is 0-12, and higher scores mean worse outcome.
Endoscopic remission | 8 weeks
  defined as Mayo endoscopic score ≤ 1
Clinical remission | 8 weeks
  overall score ≤2 [and no individual subscore >1]
Symptomatic remission | 2, 4, 6, and 8 weeks
  Stool frequence subscore = 0 (or = 1 with a ≥ 1-point decrease from baseline) and rectal bleeding subscore = 0
Fecal calprotectin | 4 and 8 weeks
  fecal sample
erythrocyte sedimentation rate | 4 and 8 weeks
  blood sample
C reactive protein | 4 and 8 weeks
  blood sample
pancreatic polypeptide | 4 and 8 weeks
  blood sample
norepinephrine | 4 and 8 weeks
  blood sample
acetyl choline | 4 and 8 weeks
  blood sample
acetyl choline | 8 weeks
  Intestinal mucosal tissue sample
alpha7 nicotinic acetylcholine receptor | 8 weeks
  Intestinal mucosal tissue sample
Inflammatory Bowel Disease Questionnaire Score | 4 and 8 weeks
  The range of Inflammatory Bowel Disease Questionnaire Score is 32-224, and higher scores mean worse outcome
Hospital Anxiety and Depression scale score | 4 and 8 weeks
  anxious depression. The range of Hospital Anxiety and Depression scale score is 0-21, and higher scores mean worse outcome.
Pittsburgh sleep quality index | 4 and 8 weeks
  The range of Pittsburgh sleep quality index is 0-21, and higher scores mean worse outcome.
autonomic profile characteristics | 4 and 8 weeks
  heart rate variability indicating sympathetic and parasympathetic activity

CONTACTS AND LOCATIONS:
Overall Officials: Kaichun Wu, Principal Investigator — Xijing Hospital
Locations (4):
- China (4):
  - Honghui hospital, Xi'an, Shaanxi
  - Second Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi
  - Tangdu Hospital, Xi'an, Shaanxi
  - Xijing Hospital, Xi'an, Shaanxi